CLINICAL TRIAL: NCT04356729
Title: A Phase II Trial of PD-L1 Therapy Combined With Anti-VEGF Therapy in Unresectable or Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elizabeth Buchbinder, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth Buchbinder, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-604
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Stage IV Melanoma; Unresectable Stage III Cutaneous Melanoma; Unresectable Stage IV Cutaneous Melanoma
Keywords: Metastatic stage III cutaneous melanoma; Metastatic stage IV cutaneous melanoma; Unresectable stage III cutaneous melanoma; Unresectable stage IV cutaneous melanoma
MeSH Terms: conditions — Melanoma | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab and Bevacizumab (Experimental): The research study procedures include screening for eligibility, study treatment including evaluations, a biopsy, and follow up visits.
  * Atezolizumab will be administered intravenously at a fixed predetermined dose every three weeks
  * Bevacizumab will be administered intravenously at a fixed predetermined dose every three weeks, with 21 consecutive days defined as a treatment cycle.
  Treatment will be administered on an outpatient basis Study treatment will continue until study doctors decide to stop therapy due to criteria which may include disease progression, adverse events or changes in condition. Participants will be followed for survival health information following treatment until the study ends, which could be approximately 5 years from start of treatment
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered intravenously at a fixed predetermined dose every three weeks ith 21 consecutive days defined as a treatment cycle.
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab will be administered intravenously at a fixed predetermined dose every three weeks, with 21 consecutive days defined as a treatment cycle.
  Other Names: Avastin; Mvasi

SUMMARY:
This research study is studying a combination of two drugs that change the immune system and tumor as a possible treatment for metastatic or unresectable stage III or IV cutaneous melanoma.

The names of the study drugs involved in this study are:

* Atezolizumab
* Bevacizumab

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility, study treatment including evaluations, a biopsy, and follow up visits.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied. The U.S. Food and Drug Administration (FDA) has not approved atezolizumab for this specific disease but it has been approved for other uses. The U.S. Food and Drug Administration (FDA) has not approved bevacizumab for this specific disease but it has been approved for other uses.

Atezolizumab and bevacizumab are types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack the cancer cells and stop the growth of cancer. Atezolizumab and bevacizumab work by stopping various molecules on cancer cells and body cells from working against the immune system's natural fight against cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed metastatic or unresectable stage III or IV cutaneous melanoma.
* PD-L1 negative staining in at least one biopsy sample.
* Age ≥ 18 years
* ECOG performance status ≤ 2 (Karnofsky ≥60%, see Appendix A)
* Participants may have received any number of prior therapies for treatment of their cutaneous melanoma, excluding prior treatment with anti-PD-L1 therapeutic antibodies or bevacizumab.
* Participants must have measurable disease per RECIST v1.1.
* Participants must have availability of a representative tumor specimen for exploratory biomarker research.
* Participants must have normal organ and marrow function as defined below:

  * lymphocyte count ≥ 500/mcL
  * absolute neutrophil count ≥ 1,500/mcL without granulocyte colony-stimulating factor support
  * platelets* ≥100,000/mcL
  * hemoglobin* ≥9 g/dL
  * serum bilirubin ≤1.5 x ULN with the following exception: participants with known Gilbert's Disease: serum bilirubin level ≤ 3x ULN
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN, with the following exceptions: Participants with documented liver metastases: AST and ALT ≤ 5 x ULN
  * alkaline phosphatase (ALP) ≤2.5 × institutional ULN, with the following exceptions:
  * participants with documented liver or bone metastases: ALP ≤ 5 x ULN
  * serum creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
  * serum albumin ≥ 2.5 g/dL
* For participants not receiving therapeutic anticoagulation: INR or aPTT ≤1.5 ULN
* Urine dipstick for proteinuria < 2+ (within 7 days prior to Cycle 1 Day 1). Participants discovered to have ≥ 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours. Note: Participants cannot be transfused to meet this criterion
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the last dose of atezolizumab, and 6 months after the last dose of bevacizumab.
* Examples of contraceptive methods with a failure rate of < 1 % per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 5 months after the last dose of atezolizumab and 6 months after the last dose of bevacizumab, to avoid exposing the embryo. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with symptomatic, untreated, or actively progressing CNS metastases will be excluded. If a participant has a known history of treated CNS lesions, they are eligible provided that all of the following criteria are met:
* Measurable disease, per RECIST v1.1, must be present outside the CNS.
* The participant has no history of intracranial hemorrhage or spinal cord hemorrhage.
* Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
* There is no evidence of interim progression between completion of CNS-directed therapy and the screening brain scan
* The participant has not received stereotactic radiotherapy within 7 days prior to initiation of study treatment or whole-brain radiotherapy within 14 days prior to initiation of study treatment.
* The participant has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted. Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan.
* History of leptomeningeal disease.
* Uncontrolled tumor-related pain.

  * NOTE: Participants requiring pain medication must be on a stable regimen at study entry.
  * Symptomatic lesions amendable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to enrollment. Participants should be recovered from the effects of radiation. There is no required minimum recovery period.
  * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to atezolizumab and/or bevacizumab.
* Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome,Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met: Rash must cover <10% of body surface area, Disease is well controlled at baseline and requires only low-potency topical corticosteroids, No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet. A radiation, methotrexate,retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Participants who test positive for HIV at time of screening are ineligible because of the increased risk of lethal infections when treated with marrow-suppressive therapy.
* Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Participants with a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening are eligible for the study.
* Active hepatitis C virus (HCV) infection, defined as a positive HCV antibody test followed by a positive HCV RNA test at screening. The HCV RNA test will be performed only for participants who have a positive HCV antibody test.
* Participants with active tuberculosis will be excluded.
* Significant cardiovascular disease, such as a New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study.
* History of other malignancy within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
* Prior allogeneic stem cell or solid organ transplantation.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study or within 5 months after the last dose of atezolizumab.
* Treatment with investigational therapy within 28 days prior to initiation of study treatment.
* Prior treatment with bevacizumab or prior PD-L1 targeted therapy.
* Treatment with systemic immunostimulatory agents (including, but not limited to,interferon and interleukin 2 [IL-2]) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to initiation of study treatment.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g. 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Patients on physiologic replacement doses of steroids less than 10mg daily prednisone equivalent are allowed. Higher replacement doses should be discussed with the overall PI to determine if patient can be included on the trial.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation.
* Known allergy or hypersensitivity to any component of the bevacizumab formulation.
* Inadequately controlled arterial hypertension (defined as systolic blood pressure [BP] > 150 mm Hg and/or diastolic BP >100 mmHg), based on an average of at least three BP readings at two or more sessions. Anti-hypertensive therapy to achieve these parameters is allowed.
* History of hypertensive crisis or hypertensive encephalopathy.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1 Day 1.
* History of hemoptysis (≥ 2.5 mL of bright red blood per episode) within 1 month prior to Cycle 1 Day 1.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Current or recent (within 10 days of Cycle 1 Day 1) use of aspirin (> 325 mg/day) or current or recent treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.
* Current or recent (within 10 days prior to Cycle 1 Day 1) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purpose (as opposed to prophylactic). Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR < 1.5 x ULN and aPTT is within normal limits (according to the institutional standards) within 14 days prior to Cycle 1 Day 1. Prophylactic use of low-molecular weight heparin (LMWH) (i.e., enoxaparin 40 mg/day) is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) is not recommended due to bleeding risk.
* History of abdominal or tracheoesophageal fistula, GI perforation, or intra-abdominal abscess within 6 months prior to Cycle 1 Day 1.
* Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure.
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
* Major surgical procedure within 4 weeks prior to Cycle 1 Day 1 or anticipation of need for a major surgical procedure during the study.
* History of intra-abdominal inflammatory process within 6 months prior to Cycle 1 Day 1, including, but not limited to, peptic ulcer disease, diverticulitis, or colitis.
* Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID).
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the last dose of atezolizumab and 6 months after the last dose of bevacizumab. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate in PD-L1 negative melanoma | 5 Years
  The primary endpoint for this study is overall response rate in PDL1 negative melanoma to combination anti-PD-L1 therapy and anti-VEGF therapy by RECIST criteria. The proportion of patients with complete response or partial response as best response to therapy will be summarized and presented with a two-sided, 90% Wald confidence interval.

SECONDARY OUTCOMES:
Overall survival | start of treatment and death from any cause up to 5 years
  Time from start of treatment to death
Time to tumor progression | up to 5 years
  Time to tumor progression (TTP) is the time interval between the dates of the start of trial treatment and first documentation of progressive disease
Duration of response | patients with objective response (confirmed CR or PR as best overall response) as the interval between dates of first documentation of objective response and first documentation of progressive disease up to 5 years
  The time-to-event endpoints will each be summarized using the method of KaplanMeier Point estimates for each endpoint will be presented with 90% confidence intervals derived using log(-log(endpoint)) methodology.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE 5. | initiation of study treatment, during study treatment, and 30 days after the last dose of study treatment or study discontinuation/termination, whichever occurs first up to 5 years
  Adverse events
Change tumor-infiltrating lymphocytes (TILs) | baseline and progression/treatment discontinuation up to 5 years
  Pre-treatment percentages of stromal infiltrating lymphocytes will be summarized descriptively for the two response groups and compared using Wilcoxon rank-sum tests.
  Changes in TILs between baseline and progression/treatment discontinuation will be calculated (post-pre) for each patient and summarized descriptivelyChanges in TILs between baseline and progression/treatment discontinuation will be calculated (post-pre) for each patient and summarized descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Buchbinder, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu